CLINICAL TRIAL: NCT05349760
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of AMB-05X in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: A Phase 2 Study to Evaluate Safety and Efficacy of AMB-05X in Subjects With Idiopathic Pulmonary Fibrosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: to focus resources on other studies
Sponsor: AmMax Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMB-053-01
Record Dates: First submitted 2022-03-31; First posted 2022-04-27 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: IPF
Keywords: Idiopathic Pulmonary Fibrosis; IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: 2:1 randomization of active to placebo
Who Masked: Participant, Investigator
Masking Description: IRT and unblinded pharmacists
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMB-05X (Experimental): AMB-05X will be administered every 4 weeks for 24 weeks (for 6 treatments in total).
  Interventions: Biological: AMB-05X
- Placebo (Placebo Comparator): Placebo will be administered every 4 weeks for 24 weeks (for 6 treatments in total).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AMB-05X — A fully human monoclonal immunoglobulin (IgG2) directed against c-fms
  Arms: AMB-05X
Drug: Placebo — Saline/D5W
  Arms: Placebo

SUMMARY:
AMB-053-01 is a randomized, placebo controlled, multicenter study which will enroll approximately 36 subjects ages 40 and older with IPF for 6 doses over a 24-week dosing period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥40 years old.
2. History of confirmed diagnosis of IPF
3. Chest HRCT at Screening
4. Subjects who are either:

   * Not being treated with approved IPF therapies (i.e., nintedanib or pirfenidone) or
   * Being treated with approved IPF therapies (i.e., nintedanib or pirfenidone)
5. Has FVC ≥45% predicted of normal AND DLCO ≥25% and ≤90% predicted
6. Has a FEV1/FVC ratio (Tiffeneau-Pinelli Index) ≥ 0.70
7. Has adequate hematologic, hepatic, and renal function

Exclusion Criteria:

1. Prior investigational drug use within 30 days or 5 half-lives
2. Presence of emphysema exceeding the extent of fibrosis
3. Active or anticipated need for lung transplant
4. Treatment with prednisone
5. Active cancer
6. Active or chronic infection with HCV, HBV, or HIV
7. Known active tuberculosis
8. History of or current immunosuppressive condition
9. IPF exacerbation within 12 weeks
10. Lower respiratory-tract infection requiring antibiotic therapy
11. Smoking
12. Other forms of interstitial lung disease
13. History of lung volume reduction surgery or lung transplant
14. Contraindications for forced expiratory maneuvers during spirometry
15. Unstable cardiac or pulmonary disease (other than IPF)
16. Fridericia-corrected QT interval (QTcF) ≥ 450 ms (men) or ≥ 470 ms (women)
17. History of drug or alcohol abuse -

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | Week 24
  Frequency and severity of reported treatment-emergent adverse events will be graded per CTCAE 5-point scale

SECONDARY OUTCOMES:
Pulmonary Function | Week 28
  Change in forced vital (FVC) capacity in liters
Pharmacodynamics via CSF1 | Week 28
  Plasma CSF1 assessment and other exploratory biomarkers
ST GEORGE'S RESPIRATORY QUESTIONNAIRE IDIOPATHIC PULMONARY FIBROSIS (SGRQ-I) | Week 28
  Change in health-related quality of life, as measured by St. George's Respiratory Questionnaire (SGRQ-I)
Cmax | Week 24
  Peak Plasma Concentration (Cmax) measurement
AUC | Week 24
  Area under the plasma concentration versus time curve (AUC) measurement

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Nguyen, MD, Study Director — AmMax Bio, Inc.

IPD SHARING:
Plan to Share IPD: No